CLINICAL TRIAL: NCT03736694
Title: A Randomized Controlled Trial to Compare the Effects of Cognitive Behavioral Therapy Workshop, Sleep Hygiene Education Workshop and Self-Help Cognitive Behavioral Therapy on Adults With Sleep Impairment in Hong Kong
Brief Title: Low-intensity Cognitive-behavioural Therapy for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chung Ka-Fai, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 18-396
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Insomnia
Keywords: Insomnia; Cognitive behavioural therapy for insomnia; Sleep hygiene education
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled trial (RCT) will be performed to compare the effectiveness of the 3 types of therapies.
  After recruitment and assessment for inclusion and exclusion criteria, the participants are randomly assigned with numbers generated by computer and divided equally into 3 groups managed by an independent administrator.
  The first intervention group (Group 1) will attend one half-day cognitive behavioural therapy for insomnia (CBTI) workshop in the community setting. The second intervention group (Group 2) will receive self-help CBTI. The control group (Group 3) will receive sleep hygiene education (SHE).
Who Masked: Investigator, Outcomes Assessor
Masking Description: After recruitment and assessment for inclusion and exclusion criteria, the participants are randomly assigned with numbers generated by computer and divided equally into 3 groups managed by an independent administrator.
  The participants are required to fill in online questionnaires themselves to prevent possible biases during outcome assessments.
  The participants will be labelled by numbers without any personal information or intervention group allocated during data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBTI Workshop (Experimental): The first intervention group (Group 1) will attend one half-day CBTI workshop in the community setting. The workshop is subdivided into 4 sessions, covering topics regarding regulation of stimuli, limit of sleeping duration, relaxation, sleep hygiene and alteration of cognitive beliefs (Arnedt, Cuddihy, & Swanson, et al, 2014; Morin, Savard, Ouellet, & Daley, 2003). One workshop has the capacity of 30 participants.
  Interventions: Behavioral: Cognitive behavioural therapy for insomnia
- Self-Help CBTI (Experimental): The second intervention group (Group 2) will receive self-help CBTI. A CBTI webpage will be set up and the subjects are asked to review all the materials in it. The content is the same as that in Group 1.
  Interventions: Behavioral: Cognitive behavioural therapy for insomnia
- SHE Workshop (Active Comparator): The control group (Group 3) will receive SHE. To ensure uniformity of the therapy model, the participants will also need to attend one half-day face-to-face session, covering topics related to sleep hygiene only. The capacity is also 30 participants.
  Interventions: Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy for insomnia — CBTI involves habitual, belief and attitude alterations so as to eliminate factors preventing sleep (Morin, Savard, Ouellet, & Daley, 2003). It is recommended by the American College of Physicians as the first-line therapy for insomnia (Qaseem, Kansagara, Forciea, Cooke, & Denberg, 2016). CBTI workshops are a relatively novel and emerging way of delivery which involves a greater number of patients than group CBTI, increases availability and accessibility by concentrating the content into half or whole day and taking place in the community settings, and reduces diagnostic labeling and cost (Bonin, Beecham, Swift, Raikundalia, & Brown, 2014; Swift, Stewart, Andiappan, Smith, Espie, & Brown, 2012). Self-help CBTI involves independent learning of the provided materials via the Internet, video or audio recording, books and pamphlets (Bruin, Bogels, Oort, & Meijer, 2015).
  Arms: CBTI Workshop; Self-Help CBTI
Behavioral: Sleep hygiene education — SHE, is commonly provided verbally or through leaflets during consultations (Espie, 2009), and is also included as a part of CBTI (Morin, Savard, Ouellet, & Daley, 2003).
  Arms: SHE Workshop

SUMMARY:
A randomized controlled trial is proposed to compare the effectiveness of workshop-based and self-Help cognitive behavioral therapy for insomnia (CBTI), and sleep hygiene education (SHE) to treat insomnia in Hong Kong adolescent and adult patients, in terms of alleviation of insomnia severity, reduction in associated insomnia symptoms/ complications, and enhancement in quality of life. Insomnia is prevalent in Hong Kong and can cause severe impacts on patients and society, but there is a dearth of related research in the local population. Therefore, it is significant to conduct this study. A total of 210 participants aged > 18 with insomnia will be recruited and randomized into 3 groups to receive one of the 3 treatments. Outcomes will be measured using relevant questionnaires filled in at the baseline, 6 and 12 weeks afterwards. The results obtained will be compared within each group and among the 3 groups using statistical testing to determine the most effective treatment option for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged 16 or above
* Satisfy the DSM-5 criteria for insomnia, i.e. inability to fall or keep asleep, or wake up too early for 3 days or more per week, throughout a minimum period of 1 month (instead of 3 months in the diagnostic criteria D) using the Brief Insomnia Questionnaire. This is to include episodic insomnia which is considered as an 'other specified insomnia disorder' in DSM-5.
* Score at least 10 points in Insomnia Severity Index
* Able to read and understand Cantonese
* Have Internet access

Exclusion Criteria:

* Suffer from recently diagnosed and untreated medical, psychiatric or sleep disorders that likely contribute to the onset and maintenance of insomnia, e.g. major depressive disorder, obstructive sleep apnea, restless legs syndrome, chronic pain.
* Currently receiving CBTI or SHE
* Work on irregular rotational shift

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia severity | Baseline assessment (Week 0); Short-term follow-up (Week 8); Long-term follow-up (Week 16)
  To identify whether CBTI workshop, self-help CBTI or SHE workshop results in the greatest alleviation of insomnia severity using the Insomnia Severity Index, which allows the patients to rate their perceived severity and satisfaction level towards their current conditions (Arnedt, Cuddihy & Swanson, et al, 2014; Wong, Zhang & Li, et al, 2017).

SECONDARY OUTCOMES:
Change in Symptoms of Mood disorders | Baseline assessment (Week 0); Short-term follow-up (Week 8); Long-term follow-up (Week 16)
  To identify which of the 3 therapies brings the largest reduction mood disorders through the Hospital Anxiety and Depression Scale.
Change in Quality of life | Baseline assessment (Week 0); Short-term follow-up (Week 8); Long-term follow-up (Week 16)
  To investigate which of the 3 therapies improves the quality of life of patients to the greatest extent using the Short-Form Six-Dimension Health Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong